CLINICAL TRIAL: NCT00187824
Title: Regulation of Endocrine, Metabolic, Immune and Bioenergetic Responses in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Other Study IDs: 04/Q0505/2
Record Dates: First submitted 2005-09-11; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2004-03

CONDITIONS: Sepsis; Critical Illness
Keywords: prospective; observational; hormonal; inflammatory; vioenergetic; immune; sepsis
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The hypothesis of this study is that bioenergetic failure in human sepsis, related to endocrine, metabolic and mitochondrial dysfunction, is a major determinant of defective host immune responses, increasing disease severity and risk of death. The objectives of this study are to examine the relationship between the severity of illness, and temporal changes in the activity of endocrine, metabolic and bioenergetic pathways, and consequent immune dysfunction in critically ill patients with sepsis and multiple organ failure in the Intensive Care Unit.

DETAILED DESCRIPTION:
The objectives of this study are to examine the relationship between the severity of illness, and temporal changes in the activity of endocrine, metabolic and bioenergetic pathways, and consequent immune dysfunction in critically ill patients with sepsis and multiple organ failure in the Intensive Care Unit.

This study will be undertaken using sequential blood sampling (until ICU discharge) and muscle biopsies (to a maximum of 5) in critically ill patients (a) with or (b) without sepsis plus a comparator group undergoing elective orthopaedic surgery. A variety of hormonal, cytokine, immune and mitochondrial measures wil lbe then made to assess whether any relationship exists between alterations in these different pathways, and whether eventual survivors and non-survivors can be distinguished.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: healthy control patients Patients undergoing elective total hip replacement will be eligible for enrollment in Group 1 after written informed consent has been obtained. Only 1 blood sample and 1 fat and muscle biopsy will be taken intra-operatively

Group 2: non-septic, critically ill patients Patients requiring intensive care within 48 hours of admission to hospital from home, for a non-septic/non-inflammatory pathology will be eligible for enrollment in the study after informed agreement has been obtained from the closest family member (see Consent below). At enrolment, Group 2 patients must have received mechanical ventilation commencing within 48 hours of admission to intensive care, should be likely to require mechanical ventilation for at least 48 hours, and must not fulfil the 2001 International Sepsis Definition Conference criteria for severe sepsis or septic shock

Group 3: patients with severe sepsis or septic shock Patients requiring intensive care within 48 hours of admission to hospital from home, and evidence of severe sepsis (organ dysfunction due to infection) or septic shock as defined by the 2001 International Sepsis Definition Conference criteria, will be eligible for enrollment in the study after informed agreement has been obtained from their next-of-kin. Patients with underlying chronic liver disease are excluded from this group, and will be enrolled separately into Group 4.

Group 4: patients with severe sepsis and underlying chronic liver disease Patients requiring intensive care admission, with underlying Child-Pugh Class A or B, biopsy-proven liver cirrhosis, within 24 h of the onset of severe sepsis (organ dysfunction due to infection) or septic shock as defined by the 2001 International Sepsis Definition Conference criteria), will be eligible for enrollment in the study after informed agreement has been obtained from their next-of-kin

Exclusion Criteria:

- Age <18 years

Child-Pugh Class C liver disease

Chronic dialysis-dependent renal failure

Hepatitis B or C infection

Immunosuppression (e.g. haematological malignancy, neutropenia, HIV infection)

Immunosuppressive drug therapy within past 6 months

Patient receiving oral or IV steroid therapy for greater than 1 week, within 6 months prior to ICU admission

Muscle biopsy contraindicated in presence of coagulopathy (INR >2, platelet count < 30,000)*

Next-of-kin declines agreement / patient declines consent

Patient receiving thyroid hormone therapy prior to ICU admission

*This does not exclude enrolment into the study, particularly in the case of Group 4 patients who frequently develop a coagulopathy as part of their underlying liver dysfunction

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-07; Study Completion 2007-08

CONTACTS AND LOCATIONS:
Overall Officials: Mervyn Singer, MBBS MD FRCP, Study Director — UCL/UCLH; Geoff Bellingan, PhD FRCP, Principal Investigator — UCL/UCLH; Paul Glynne, PhD FRCP, Principal Investigator — UCL/UCLH
Locations (1):
- UCL Hospitals NHS Foundation Trust, London, London, United Kingdom

REFERENCES:
- [Derived] Carre JE, Orban JC, Re L, Felsmann K, Iffert W, Bauer M, Suliman HB, Piantadosi CA, Mayhew TM, Breen P, Stotz M, Singer M. Survival in critical illness is associated with early activation of mitochondrial biogenesis. Am J Respir Crit Care Med. 2010 Sep 15;182(6):745-51. doi: 10.1164/rccm.201003-0326OC. Epub 2010 Jun 10. PMID 20538956